CLINICAL TRIAL: NCT00815854
Title: Folate Pharmacogenomics and Risk of Atypical Antipsychotic Metabolic Side Effects
Brief Title: Examining Risk Factors for Atypical Antipsychotic Metabolic Side Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Vicki Ellingrod, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: R01MH082784 (NIH); R01MH082784 (NIH); R01MH082784-01 (NIH); DATR A5-ETSE
Record Dates: First submitted 2008-12-29; First posted 2008-12-31 (Estimated); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Schizophrenia
Keywords: Antipsychotic; Metabolic Syndrome; Insulin Resistance; Endothelial Function
MeSH Terms: conditions — Schizophrenia; Metabolic Syndrome; Insulin Resistance | interventions — Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Folate (Experimental): During Phase 1, participants will undergo screening for metabolic syndrome and have genetic makeup, body size, and endothelial functioning measured. During Phase 2, participants will receive daily folic acid as a treatment for metabolic syndrome.
  Phase 2B participants will receive either daily folic acid or placebo as a treatment for metabolic syndrome.
  Interventions: Dietary Supplement: Folic Acid
- Placebo (Placebo Comparator): During Phase 1, participants will undergo screening for metabolic syndrome and have genetic makeup, body size, and endothelial functioning measured. During Phase 2, participants will receive daily folic acid as a treatment for metabolic syndrome.
  Phase 2B participants will receive either daily folic acid or placebo as a treatment for metabolic syndrome.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Folic Acid — 5 mg of folic acid taken daily for 3 months in an open label fashion
  Other Names: Folate
  Arms: Folate
Other: Placebo — Subjects may receive placebo (a sugar pill) for 4 months
  Arms: Placebo

SUMMARY:
This study will examine possible causes of metabolic side effects in people taking atypical antipsychotic (AAP) medications.

DETAILED DESCRIPTION:
Antipsychotic medications are used to treat some of the most severe symptoms of mental illness, such as hallucinations and irrational outbursts. Atypical antipsychotics (AAPs) are a group of newer, second generation antipsychotic medications that effectively treat psychotic symptoms but that also have severe side effects. One side effect is an increased risk of metabolic syndrome, which is a cluster of conditions that together increase the risk of heart disease, stroke, type 2 diabetes, and endothelial dysfunction-dysfunction of the cells that line the inner surface of blood cells. Schizophrenic patients taking atypical antipsychotics are more than twice as likely as the general population to experience metabolic syndrome. Certain genetic variants associated with folate metabolism, as well as low dietary folate, may lead to the development of metabolic syndrome and its associated diseases. These factors have been studied in the general population, but not in a group of schizophrenic patients taking antipsychotics. This study will examine the relationship among folic acid, variants in the gene methylenetetrahydrofolate reductase, and metabolic syndrome and its associated diseases in people with schizophrenia who are taking atypical antipsychotics. The study will also evaluate the use of folic acid supplementation for treating metabolic syndrome in this population.

Participation in this study will involve two phases. The first phase will involve recruitment, screening, and testing of participants taking antipsychotics and will last 4 years. During this phase, participants will attend one study visit in which they will undergo a screening for metabolic syndrome and have the following measured: endothelial functioning, body size, diet, physical activity, medication history, and genetic makeup. Participants who have metabolic syndrome will be invited to participate in Phase 2.

Phase 2 will run concurrently with Phase 1, but will extend to 5 years, in order to give all participants an opportunity to continue from one phase to the next if they meet entry criteria. Participants in Phase 2 will attend four study visits over the course of 3 months: one at the beginning of the phase and one after each month of the study. After the first study visit, participants will be given folic acid to take daily for the 3 months. At each study visit, participants will be asked about thoughts, illness, functioning, diet, medication side effects, recent medication history, smoking history, alcohol intake, and exercise habits. On the first and last visits, participants will undergo additional tests of genetics, blood hormone levels, and blood vessel functioning, and additional measurements will be made of height, weight, vital signs, and body size. The Phase 2 study is now inactive.

Phase 2B is active and currently recruiting participants. This is a randomized, placebo controlled study of folate supplementation. Participants in phase 2B will attend 6 study visits over the course of 6 months. At the first study visit they will be randomized to either folic acid 5mg daily for 4 months or placebo. This 4 month period is followed by a 2 month follow up visit, when no supplementation is given. At each study visit, participants will be asked about thoughts, illness, functioning, diet, medication side effects, recent medication history, smoking history, alcohol intake, and exercise habits. On the first and last visits, participants will undergo additional tests of genetics, blood hormone levels, and blood vessel functioning, and additional measurements will be made of height, weight, vital signs, and body size.

ELIGIBILITY:
Inclusion Criteria for Phase 1:

* DSM-IV diagnosis of schizophrenia, schizophreniform disorder, schizoaffective disorder, or psychosis not otherwise specified
* Treatment with one of the following atypical antipsychotics (AAPs) for at least 6 months: clozapine, olanzapine, risperidone, quetiapine, aripiprazole, or ziprasidone

Inclusion Criteria for Phase 2:

* Previous participation in Phase 1 pharmacogenomic study
* Meets metabolic syndrome criteria
* No medication changes for 6 months, including antipsychotic medication changes and changes in any other medications related to treating metabolic syndrome, diabetes, hypertension, or hyperlipidemia

Exclusion Criteria for Phases 1 and 2:

* Presence of any serious medical condition that would significantly affect weight changes, such as neoplastic or thyroid disease
* Diagnosis of active substance dependence or use of illicit substances within the past month
* History of type 2 diabetes mellitus prior to AAP use
* Past history of or currently has pernicious, aplastic, or normocytic anemia with a B12 deficiency

Inclusion criteria for Phase 2B:

* At least 18 years old and presence of a DSM-IV diagnosis of schizophrenia, schizophreniform disorder, schizoaffective disorder, or psychosis NOS
* Receiving atypical antipsychotic medication for at least 6 months
* Currently meet ≥ 2 of the NCEP-ATP-III criteria for metabolic syndrome
* No medication changes within the last two months
* Vitamin B12 levels within normal laboratory levels
* No illicit drug use in the past month

Exclusion Criteria for Phase 2B

* Inability to give informed consent or unwillingness to participate
* Presence of any serious medical conditions that would significantly affect weight changes (i.e. neoplastic or uncontrolled thyroid disease)
* Blood pressure lower than 90/60 mmHg
* History of Type 2 Diabetes Mellitus prior to AAP use
* History of hypersensitivity or allergic reaction to folic acid or any of the product ingredients
* Current pregnancy or nursing
* Current substance dependence diagnosis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2008-10; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Endothelial functioning | Measured at baseline and after 3 months, and then at a two month follow up visit
  Using the EndoPAT machine (Itamar) we will measure the Reactive hyperemia index (RHI)

SECONDARY OUTCOMES:
metabolic syndrome | measured at baseline, endpoint, and follow up
  Metabolic Syndrome is defined as having any 3 of the following: 1) abdominal obesity characterized by waist circumference of >40 inches for men or >35 inches for women, 2) triglycerides ≥150 mg/dL, 3) HDL cholesterol <40 mg/dL for men and <50 mg/dL for women or receiving a lipid lowering agent), 4) blood pressure ≥130/≥85 mmHg or treatment for hypertension, or 5) fasting glucose ≥100 mg/dL or treatment of diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Vicki L. Ellingrod, PharmD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States